CLINICAL TRIAL: NCT02672605
Title: Measurement of Individual-Level Abortion Stigma Resulting From Pennsylvania State-Mandated Abortion Consent Language: A Pilot Randomized Controlled Trial
Brief Title: Measurement of Individual Level of Abortion Stigma Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 823273
Record Dates: First submitted 2016-01-26; First posted 2016-02-03 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2016-07

CONDITIONS: Abortion Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Participant completes a survey measuring abortion stigma prior to receiving the mandatory Pennsylvania State consent for their abortion.
- Investigational (Experimental): Participant completes a survey measuring abortion stigma after receiving the mandatory Pennsylvania State consent for their abortion.
  Interventions: Other: Pennsylvania State Abortion Consent

INTERVENTIONS:
Other: Pennsylvania State Abortion Consent — Measuring the level of stigma felt pre- or post-exposure to the abortion consent language.
  Arms: Investigational

SUMMARY:
This study is a randomized controlled trial designed to measure abortion stigma related to the Pennsylvania Abortion Control Act. Women seeking abortion will be randomized to receive the validated Individual Level Abortion Stigma Scale either before or after consent via the Pennsylvania Abortion Control Act language. The primary outcome will be the stigma scores in the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. Women ≥18 years old
2. Seeking induced abortion for any indication
3. Gestation ≤ 24 weeks
4. Plan for procedural or state consent at current visit
5. Willing and able to consent in English

Exclusion Criteria:

1. Have previously been consented in the current pregnancy using the Pennsylvania Abortion Control Act consent language
2. Have previously had an abortion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Individual level stigma scores | Stigma store is collected during one 30-minute study visit, either directly prior or directly following the patient being consented using the PA Abortion Control Act language

CONTACTS AND LOCATIONS:
Overall Officials: Sarita Sonalkar, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Family Planning and Pregnancy Loss Center, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No